CLINICAL TRIAL: NCT00003334
Title: Phase II Study of Doxil and Paclitaxel in Patients With Endometrial, Tubal, and Sarcomas of Gynecologic Origin
Brief Title: Combination Chemotherapy in Treating Patients With Endometrial Cancer, Fallopian Tube Cancer, or Sarcoma of the Female Reproductive Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066300; NYU-9708; NYGOG-NY9708; NCI-G98-1427
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Sarcoma
Keywords: stage IV endometrial carcinoma; recurrent endometrial carcinoma; fallopian tube cancer; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma; ovarian sarcoma; ovarian carcinosarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma; Sarcoma, Endometrial Stromal | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining doxorubicin and paclitaxel in treating patients who have recurrent or refractory endometrial cancer, fallopian tube cancer, or sarcoma of the female reproductive tract.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response to doxorubicin HCl liposome and paclitaxel in patients with endometrial cancer, tubal cancers, and sarcomas and carcinosarcomas (mixed mesodermal tumors) of gynecologic origin. II. Define the safety profile of the combination of doxorubicin HCl liposome and paclitaxel in this patient population.

OUTLINE: Patients are stratified into two groups. Group 1 consists of patients with untreated endometrial and tubal cancers and Group 2 consists of patients with sarcomas and carcinosarcomas (mixed mesodermal tumors) of gynecologic origin subdivided into no or prior therapy. Patients receive doxorubicin HCl liposome intravenously on day 1 of each treatment course. Paclitaxel is administered intravenously weekly on days 1, 8, and 15 of each course. Courses are repeated every 21 days. Treatment continues in the absence of unacceptable toxic effects or disease progression. Patients are followed every 3 months for 2 years, then every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 28-60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed recurrent or refractory carcinoma of the endometrium or fallopian tubes or sarcomas of gynecologic origin including mixed mesodermal sarcomas Documented recurrence or persistence of disease after appropriate surgical and/or radiation therapy Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Platelet count at least 50,000/mm3 Granulocyte count at least 1,000/mm3 Hepatic: SGOT and SGPT no greater than 3 times upper limit of normal (ULN) Bilirubin no greater than 3 times ULN Renal: Creatinine less than 2.5 mg/dL Cardiovascular: MUGA at least lower limit of normal Normal ejection fraction and/or stable cardiac status Other: No medical or social factors that would interfere with compliance Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No serious concurrent illness requiring immediate therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 months since prior combined modality or adjuvant chemotherapy Prior doxorubicin allowed if cumulative dose is recorded Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: Not specified Other: At least 30 days since prior noncytotoxic experimental antiemetic or antifungal investigational drugs

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-03; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (5):
- United States (5):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York

REFERENCES:
- [Result] Hornreich G, Muggia FM, Wadler S, et al.: Phase II combination doxil-paclitaxel (PacliDox) in uterine carcinomas and sarcomas - an active regimen: a New York Gynecologic Oncology Group study. [Abstract] Society of Gynecologic Oncologists 2003 Annual Meeting on Women's Cancer, January 31 - February 2, 2003, New Orleans, Louisiana. A-606, 2003.